CLINICAL TRIAL: NCT02710708
Title: Single-arm, Open-label, Interventional Study to Observe the Safety and Efficacy Profile of the Combined Oral Contraceptive YAZ®, a 24-day Cyclic Regimen Containing Drospirenone 3 mg and Ethinyl Estradiol 20 µg During a Treatment Duration of 6 Cycles: a Post-authorization Safety and Efficacy Study in Chinese Women
Brief Title: YAZ Post Authorization Safety Study (PASS)/Post Authorization Efficacy Study (PAES) in China
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18261
Record Dates: First submitted 2016-03-14; First posted 2016-03-17 (Estimated); Last update posted 2019-06-28 (Actual); Status verified 2019-06

CONDITIONS: Contraception
Keywords: birth control,; contraceptives safety,; contraceptives efficacy,; moderate acne vulgaris
MeSH Terms: interventions — drospirenone and ethinyl estradiol combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ethinyl Estradiol 20 (EE20)/DRSP (YAZ, BAY86-5300) (Experimental): Chinese women between 18 and 45 years old inclusive (smokers not older than 35 years old) requesting oral contraception who have no contraindication to YAZ will be recruited for the study. Women who underwent surgical or medical abortions will also be recruited.
  Interventions: Drug: EE20/DRSP (YAZ, BAY86-5300)

INTERVENTIONS:
Drug: EE20/DRSP (YAZ, BAY86-5300) — YAZ (DRSP 3 mg/EE 20 µg), oral route, 6 cycles of 28 days per cycle, each cycle comprising 24 days of active tablets followed by 4 days of placebo tablets

SUMMARY:
The primary objective is to assess the safety profile of YAZ in Chinese women, including adverse drug reactions (ADRs).

The secondary objectives are to investigate the rate of unintended pregnancies, the cycle control for subjects with and without preceding abortion, the bleeding pattern of subjects with and without preceding abortion (including the abortion-related bleeding pattern) and the efficacy in moderate acne vulgaris.

Another objective is to investigate the effect on dysmenorrhea.

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated informed consent
* Chinese female subjects requesting oral contraception, including subjects who underwent abortion (medical or surgical)
* Planned use of combined oral contraceptives for at least 6 cycles
* Age: 18 to 45 years (inclusive); smokers must not be older than 35 years at the time of informed consent
* At least 4 weeks postpartum for women who are not breastfeeding or after a second trimester abortion

Exclusion Criteria:

* Evidence or suspicion of incomplete abortion (medical abortion subjects must have complete abortion confirmed by ultrasound [endometrial thickness ≤ 15 mm]).
* Pregnancy or lactation
* Menstrual disorders consistent with ovarian failure (eg, oligomenorrhea, amenorrhea, hypomenorrhea)
* Abuse of alcohol, drugs, or medicine (eg, laxatives)
* Inability to cooperate with the study procedures for any reason (eg, language comprehension, psychiatric illness, inability to get to the study site).
* Any diseases or conditions that can compromise the function of body systems and could result in altered absorption, excessive accumulation, impaired metabolism, or altered excretion of the study medication
* Any diseases or conditions that might interfere with the conduct of the study or the interpretation of the results
* Any contraindication to YAZ according to the Chinese label, such as:

  * Renal impairment
  * Adrenal insufficiency
  * A high risk of arterial or venous thromboembolic diseases. Examples include subjects who are known to:

    * Have deep vein thrombosis or pulmonary embolism, now or in the past
    * Have cerebrovascular disease
    * Have coronary artery disease
    * Have thrombogenic valvular or thrombogenic rhythm diseases of the heart (eg, subacute bacterial endocarditis with valvular disease, or atrial fibrillation)
    * Have inherited or acquired hypercoagulopathies
    * Have uncontrolled hypertension
    * Have diabetes mellitus with vascular disease
    * Have headaches with focal neurological symptoms or have migraine headaches with or without aura if over age 35
  * Breast cancer or other estrogen- or progestin-sensitive cancer, now or in the past
  * Liver tumors, benign or malignant, or liver disease
* Hypersensitivity to any ingredient of the study drug
* Undiagnosed abnormal genital bleeding
* Sterilized subjects or concomitant use of other hormonal contraception, intrauterine device (IUD), or intrauterine system (IUS) during the study
* For subjects qualifying for the moderate acne subgroup:

  * Subjects with acne and atopy, comedonal acne or acne conglobata, sandpaper acne or acne with multiple large nodes, cysts, fistular comedones, or abscessing fistular ducts
  * Use of preparations that have an acne-inducing effect (eg, iodinated or bromated drugs, tuberculostatics, lithium, vitamin B1 [>1.5 mg daily], B6 [>2 mg daily], B12 [>6 µg daily], corticoids, adrenocorticotropic hormone anabolics, quinine, disulfiram, methoxypsoralene, phenobarbital, phenytoin, trimethadione, thyroid depressants, and certain oily cosmetics)
  * Subjects undergoing systemic acne treatment

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1921 (Actual)
Dates: Start 2016-05-27 (Actual); Primary Completion 2018-07-03 (Actual); Study Completion 2018-07-03 (Actual)

PRIMARY OUTCOMES:
Number of subjects with adverse drug reactions (ADRs) | 6 months

SECONDARY OUTCOMES:
Number of unintended pregnancies as measured by the Pearl Index (PI) | 6 months
Cycle control for subjects with and without proceeding abortion | 6 months
Number of bleeding days | Up to 90 days.
Number of bleeding episodes | Up to 90 days.
Number of Acne lesions | 6 months

OTHER OUTCOMES:
Severity of pain during menstruation measured by visual analog scale (VAS) | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (25):
- China (25):
  - Xiamen, Fujian
  - Guangzhou, Guangdong
  - Shenzhen, Guangdong
  - Liuchow, Guangxi
  - Nanning, Guangxi
  - Shijiazhuang, Hebei
  - Changshacun, Henan
  - Wuhan, Hubei
  - Yueyang, Hunan
  - Changzhou, Jiangsu
  - Nanjing, Jiangsu
  - Wuxi, Jiangsu
  - Nanchang, Jiangxi
  - Xi'an, Shaanxi
  - Weifang, Shandong
  - Zibo, Shandong
  - Taiyuan, Shanxi
  - Chengdu, Sichuan
  - Ürümqi, Xinjiang
  - Kunming, Yunnan
  - Hangzhou, Zhejiang
  - Wenzhou, Zhejiang
  - Beijing
  - Shanghai
  - Tianjin

REFERENCES:
- [Derived] Sun X, Qian F, He Y, Gu X, Di W. Safety and Efficacy of Combined Oral Contraceptive Ethinyl Estradiol/Drospirenone (YAZ) in Chinese Women: A Single-Arm, Open-Label, Multicenter, Post-Authorization Study. Adv Ther. 2020 Feb;37(2):906-917. doi: 10.1007/s12325-019-01210-2. Epub 2020 Jan 16. PMID 31950432